CLINICAL TRIAL: NCT03601286
Title: Phase I/II Study of Lentiviral Gene Transfer for SCID-X1 With Low Dose Targeted Busulfan
Brief Title: Lentiviral Gene Therapy for X-linked Severe Combined Immunodeficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16IC17
Record Dates: First submitted 2018-02-22; First posted 2018-07-26 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Severe Combined Immunodeficiency, X-Linked
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lentiviral vector transduced CD34+ cells (Experimental): Single arm, non-randomised cohort of up to 5 patients with X-linked Severe Combined Immunodeficiency. CD34+ cells will be collected via bone marrow harvest or leukapheresis. The collected cells will then be purified, cultured and transduced with the G2SCID lentiviral vector. Transduced cells will be frozen. A minimum of 2.5 x 106/kg CD34+ cells after transduction with a minimum transduction efficiency of 0.7 copies/cell is required for infusion into the patient. The patient will receive non-myeloablative conditioning with intravenous busulfan the two or three days prior to cell infusion. The frozen cells will be thawed on the day of infusion and the cells administered according to hospital procedures. The patient will remain in hospital until sufficient cover of the patient's immune system
  Interventions: Drug: Lentiviral vector transduced CD34+ cells

INTERVENTIONS:
Drug: Lentiviral vector transduced CD34+ cells — Gene therapy for X-linked Severe Combined Immunodeficiency will be performed by introduction a normal copy of the IL2RG gene into the blood forming stem cells (CD34+ cells) of the patient's bone marrow by using a type of gene delivery system (in this trial called a lentiviral vector). The gene corrected cells are then transplanted back into the patient.
  Other Names: G2SCID lentiviral vector transduced CD34+ cells

SUMMARY:
Severe combined immunodeficiency disorder (SCID) is a heterogeneous group of inherited disorders characterized by a profound reduction or absence of T lymphocyte function, resulting in lack of both cellular and humoral immunity. SCID arises from a variety of molecular defects which affect lymphocyte development and function. The most common form of SCID is an X-linked form (SCID-X1), which accounts for 30-50% of all cases. SCID-X1 is caused by defects in the common cytokine receptor gamma chain, which was originally identified as a component of the high affinity interleukin-2 receptor (IL2RG).

Allogeneic haematopoietic stem cell transplantation (HSCT), which replaces the patient's bone marrow with that of a healthy donor, is the only treatment that definitively restores the normal function of the bone marrow. HSCT is the first choice of treatment for patients with signs of bone marrow failure and a fully-matched related donor. However, patients without a fully-matched related donor have much worse overall outcomes from HSCT.

This study will investigate whether patients with SCID-X1 without a fully matched related donor may benefit from gene therapy. To do this the investigators propose to perform a phase I/II clinical trial to evaluate the safety and efficacy (effect) of gene therapy for SCID-X1 patients using a lentivirus delivery system containing the IL2RG gene. Up to 5 eligible SCID-X1 patients will undergo mobilisation and harvest of their haematopoietic stem precursor cells (HPSCs). In the laboratory the disabled lentivirus will be used to insert a normal human IL2RG gene into the patient's harvested HPSCs. Patients will receive chemotherapy conditioning prior to cell infusion, in order to enhance grafting. The genetically corrected stem cells will then be re-infused into the patient. Patients will be followed up for 2 years. This trial will determine whether gene therapy for SCID-X1 using a lentiviral vector is safe, feasible and effective

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SCID-X1 based on immunophenotype and lack of T cell function (proliferation to PHA <10% of the lower limit of normal for the laboratory) AND confirmed by a mutation in IL2RG
2. Lack of an HLA identical (A, B, C, DR, DQ) related donor
3. Age <5 years
4. Signed informed consent
5. Documentation of willingness to follow up for 15 years post-infusion
6. If the patient has previously undergone allogeneic transplant or gene therapy, insufficiency of graft-derived T cell engraftment must be documented.
7. Age at least 8 weeks of age by the time of busulfan administration

Exclusion Criteria:

1. Patients with an active, therapy-resistant infection. Infections that are known to be highly morbid in SCID patients will be considered active and therapy-resistant if the infectious agent is repeatedly isolated despite a minimum of 2 weeks of appropriate therapy and is associated with significant organ dysfunction (including but not limited to abnormalities listed below).

   1. Mechanical ventilation including continuous positive airway pressure
   2. Abnormal liver function defined by AST and ALT >10 times the upper range of normal OR Bilirubin >2 mg/dL
   3. Shortening fraction on echocardiogram <25% or ejection fraction <50%
   4. Renal failure defined as glomerular filtration rate <30 ml/min/1.73 m2 or dialysis dependence
2. Uncontrolled seizure disorder
3. Encephalopathy
4. Documented coexistence of any disorder known to affect DNA repair
5. Diagnosis of active malignant disease other than EBV-associated lymphoproliferative disease
6. Patients with evidence of infection with HIV-1
7. Previous allogeneic transplant with cytoreductive chemotherapy
8. Major (life-threatening) congenital anomalies. Examples of "major (life-threatening) congenital anomalies" include, but are not limited to: unrepaired cyanotic heart disease, hypoplastic lungs, anencephaly or other major central nervous system malformations, other severe non-repairable malformations of the gastrointestinal or genitourinary tracts that significantly impair organ function.
9. Other conditions which in the opinion of the P.I. or Co-investigators, contra-indicate collection and/or infusion of transduced cells or indicate patient's inability to follow the protocol. These may include for example clinical ineligibility to receive anaesthesia, severe deterioration of clinical condition of the patient after collection of bone marrow but before infusion of transduced cells, or documented refusal or inability of the family to return for scheduled visits. There may be other unforeseen rare circumstances that would result in exclusion of the patient, such as sudden loss of legal guardianship.

Ages: 8 Weeks to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — As SCID-X1 is an X-linked disorder, women/girls will not be enrolled.
Enrollment: 5 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Measure event-free survival after 1 year after gene transfer | 1 year
  Event-free survival at 1 year post-infusion. Events will include death, infusion of unmanipulated back-up product for failure of haematopoietic recovery, and allogeneic transplant performed for poor immune reconstitution
Measure T cell immune reconstitution: CD3+ T cell count | 1 year
  T cell reconstitution at 1 year post-infusion: CD3+ T cell count ≥300 cells/microliter in peripheral blood
Measure T cell immune reconstitution; gene marking | 1 year
  T cell reconstitution at 1 year post-infusion: Gene marking ≥0.1 copies/cell in sorted CD3+ T cells

SECONDARY OUTCOMES:
Measure overall survival | 2 years
  Measure overall survival at 2 years post-infusion
Measure event-free survival | 2 years
  Measure event-free survival at 2 years post-infusion
Incidence of adverse events related to gene therapy | up to 2 years post-infusion of gene therapy
  Incidence of adverse events related to gene therapy
Enumeration of absolute lymphocyte count determined by routine complete reconstitution | up to 2 years post-infusion of gene therapy
  Enumeration of absolute lymphocyte count determined by routine complete blood counts (CBC)
Haematopoietic recovery after receipt of busulfan | up to 6 weeks post-infusion of gene therapy
  Haematopoietic recovery is defined as absolute neutrophil count above 0.5 x10^9 /l for three consecutive days, achieved within 6 weeks following infusion.
Measure absolute numbers of T, B and NK lymphocytes | up to 2 years post-infusion of gene therapy
  Absolute numbers of T, B and NK lymphocytes
Calculate percentage of naïve and memory T cell subsets | up to 2 years post-infusion of gene therapy
  Percentage of naïve and memory T cell subsets
Measure laboratory results which correlates with efficacious immune reconstitution | up to 2 years post-infusion of gene therapy
  Percentage of naïve and memory B cell subsets
Determine Freedom from immunoglobulin substitution for at least 9 months | 2 years post-infusion of gene therapy
  Freedom from immunoglobulin substitution for at least 9 months
Measure serum immunoglobulin levels reconstitution | up to 2 years post-infusion of gene therapy
  Serum immunoglobulin levels
Measure proliferation of lymphocytes to phytohaemagglutinin determined by titrated thymidine incorporation reconstitution | up to 2 years post-infusion of gene therapy
  Proliferation of lymphocytes to phytohaemagglutinin determined by titrated thymidine incorporation
Measure antigen specific antibody titres to tetanus toxoid reconstitution | up to 2 years post-infusion of gene therapy
  Measure antigen specific antibody titres to tetanus toxoid
Measure T cell receptor excision circles (TREC) | up to 2 years post-infusion of gene therapy
  Measure T cell receptor excision circles (TREC)
Measure T cell receptor Vb family usage | up to 2 years post-infusion of gene therapy
  Measure T cell receptor Vb family usage
To assess the efficacy of stem cell transduction/engraftment by measuring the frequency of gene marking in peripheral blood cells | up to 2 years post-infusion of gene therapy
  Gene marking in specific lineages of peripheral blood cells. Genomic DNA isolated from each population will be assayed for VCN by quantitative PCR (qPCR). The results will be aggregated to determine the effectiveness of gene marking in the peripheral blood cells.
Measure clonal diversity of vector integrants | up to 2 years post-infusion of gene therapy
  Clonal diversity will be quantitated and used to estimate the number of transduced haematopoietic stem cells that have engrafted in the subjects. Number of sequence reads and unique integration sites will be assessed to quantify population clone diversity, distribution of integration sites and relative abundance.

OTHER OUTCOMES:
Correlation of potential biomarkers of humoral immune reconstitution with freedom from intravenous immunoglobulin substitution and antibody response to tetanus at 2 years post infusion including: Gene marking in B cells and B cell phenotype. | at 6 month, 12 month and 2 years post-infusion of gene therapy
  Correlation of potential biomarkers of humoral immune reconstitution at 6 months, 1 year, 2 years post infusion with freedom from intravenous immunoglobulin substitution and antibody response to tetanus at 2 years post infusion including: Gene marking in B cells and B cell phenotype.
Correlation of busulfan area-under-the-curve measurements prior to infusion with freedom from intravenous immunoglobulin substitution and antibody response to tetanus at 2 years post-infusion and other markers of humoral immune reconstitution | 2 years post-infusion of gene therapy
  Correlation of busulfan area-under-the-curve measurements prior to infusion with freedom from intravenous immunoglobulin substitution and antibody response to tetanus at 2 years post-infusion and other markers of humoral immune reconstitution
Evidence of insertion site sharing between 2 or more lineages at 1 year and 2 years post infusion | 1 year and 2 years post infusion of gene therapy
  Evidence of insertion site sharing between 2 or more lineages at 1 year and 2 years post infusion
Correlation of gene marking and insertion site sharing in expanded peripheral blood CD34+ cells with peripheral blood mature cell samples at 1 year and 2 years post infusion | 1 year and 2 years post infusion of gene therapy
  Correlation of gene marking and insertion site sharing in expanded peripheral blood CD34+ cells with peripheral blood mature cell samples at 1 year and 2 years post infusion
Description of T cell receptor and B cell receptor repertoire before and after infusion | Pre-harvest, 3 month, 6 month, 12 month and 2 years post infusion of gene therapy
  Description of T cell receptor and B cell receptor repertoire before and after infusion
Description of NK cell function and phenotype before and after infusion | Pre-harvest, 3 month, 6 month, 12 month and 2 years post infusion of gene therapy
  Description of NK cell function and phenotype before and after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Claire Booth, Dr, Principal Investigator — UCL Great Ormond Street Institute of Child Health; Adrian Thrasher, Prof, Principal Investigator — UCL Great Ormond Street Institute of Child Health
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No